CLINICAL TRIAL: NCT06912711
Title: Toripalimab Combined With Nimotuzumab Induction and Adjuvant Therapy for Resectable Local Recurrent Nasopharyngeal Carcinoma：A Single-arm, Phase II Clinical Tria
Brief Title: TN Induction and Adjuvant Therapy for Resectable Local Recurrent Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, YiJun Hua, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-320-NPC
Record Dates: First submitted 2025-04-03; First posted 2025-04-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; nimotuzumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Toripalimab Combined With Nimotuzumab Induction therapy then surgery and Toripalimab Combined With Nimotuzumab adjuvant Therapy
  Interventions: Drug: Toripalimab; Drug: Nimotuzumab; Procedure: surgery

INTERVENTIONS:
Drug: Toripalimab — Triplizumab (240mg, Q3W, 2 cycles, induction)and (240mg, Q3W, 15 cycles, adjuvant)
Drug: Nimotuzumab — Triplizumab (200mg, Q3W, 2 cycles, induction) and (200mg, Q3W, 15 cycles, adjuvant)
Procedure: surgery — The complete resection of the nasopharyngeal tumor and its adequate safety boundary must be performed under general anesthesia and under the guidance of nasal endoscopy through bilateral nasal passages. The anterior incisal margin should reach 1-2cm in front of the posterior column of the nasal septum, and the upper incisal margin should reach about 0.5-1cm in front of the upper margin of the posterior nostril. The lateral incisal margin and the lower incisal margin should be individually designed according to the size and location of the tumor. A safe incisal margin of 0.5-1.0cm was obtained, and then the tumor tissue and normal tissue of the incisal margin were ablated layer by layer from the upper incisal margin to the lower incisal margin until no obvious tumor remained under the naked eye.

SUMMARY:
Investigators target recurrent nasopharyngeal carcinoma that can be resected surgically: rT1, rT2 (tumor confined to the surface of the parapharyngeal space, greater than 0.5cm from the internal carotid artery), rT3 (confined to the floor of the sphenoid sinus, greater than 0.5cm from the internal carotid artery/cavernous sinus) (AJCC 8th stage), A single-arm, phase II clinical trial was designed to investigate the efficacy and safety of triplizumab combined with nituzumab in induction and adjuvant treatment of operable local recurrent nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Investigators target recurrent nasopharyngeal carcinoma that can be resected surgically: rT1, rT2 (tumor confined to the surface of the parapharyngeal space, greater than 0.5cm from the internal carotid artery), rT3 (confined to the floor of the sphenoid sinus, greater than 0.5cm from the internal carotid artery/cavernous sinus) (AJCC 8th stage), A single-arm, phase II clinical trial was designed to investigate the efficacy and safety of triplizumab combined with nituzumab in induction and adjuvant treatment of operable local recurrent nasopharyngeal carcinoma. The investigators focus on the 2-year PFS as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in and sign the informed consent in person. 2. Aged 18-65 years, male or non-pregnant female. 3. Histologically and/or cytologically confirmed recurrent nasopharyngeal carcinoma (keratinized or non-keratinized carcinoma; Differentiated or undifferentiated) 4. Patients with recurrence time more than 6 months from the end of radiotherapy; 5. Recurrent nasopharyngeal carcinoma that can be resectable: rT1, rT2 (the tumor is confined to the surface of the parapharyngeal space, and the distance from the internal carotid artery is greater than that from the internal carotid artery 0.5cm), rT3 (confined to the floor wall of the sphenoid sinus, greater than 0.5cm from the internal carotid artery/cavernous sinus) (AJCC 8th stage).

If the tumor invades the internal carotid artery, or is less than 0.5cm away from the internal carotid artery, but the invasion scope does not exceed the external edge of the internal carotid artery, it can be advanced Internal carotid artery preconditioning (including internal carotid artery embolization or stent implantation) was followed.

6. ECOG score 0-1, no serious dysfunction of heart, lung, liver, kidney and other vital organs.

7. Hemoglobin (HGB) ≥90 g/L, white blood cells (WBC) ≥4.0×109 /L, platelets (PLT) ≥100×109 /L.

8. Liver function: ALT and AST< 2.5 times the upper limit of normal (ULN), total bilirubin <2.0×ULN.

9. Renal function: serum creatinine <1.5×ULN.

Exclusion Criteria:

* 1. The pathological findings were keratinized squamous cell carcinoma (WHO type I).

  2. Received systemic or local glucocorticoid therapy within 4 weeks before enrollment.

  3. Patients who have participated in other drug clinical trials within 3 months before treatment.

  4. Patients with a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 5. Idiopathic pulmonary fibrosis, drug-induced pneumonia, institutional pneumonia (i.e., bronchiolitis obliterans), clinical symptoms or Radiation pneumonia, active pneumonia, or other moderate to severe lung disease requiring steroid treatment 6. Have a comorbiditis that requires prolonged treatment with immunosuppressive drugs or systemic or local use of immunosuppressive doses of corticosteroids.

  7. The subject has any active autoimmune disease or history of autoimmune disease (including, but not limited to, interstitial disease) Pneumonia, uveitis, enteritis, hepatitis, pituitaritis, nephritis, hyperthyroidism, hypothyroidism; Suffer from Patients with vitiligo or asthma that had completely resolved in childhood and did not require any intervention in adulthood were included; Need bronchus Dilators for medical intervention in asthma were not included).

  8. Positive HBV DNA copy number was detected in both HIV-positive and HBsAg positive patients (quantitative detection ≥ 1000cps/ml); Chronic hepatitis C blood screening positive (HCV antibody positive) with HCV RNA positive detection.

  9. Received any anti-infection vaccine (such as influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment.

  10. Pregnancy test positive women of childbearing age and breastfeeding women. 11. Patients who cannot cooperate with regular follow-up due to psychological, social, family and geographical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2029-04-20 (Estimated); Study Completion 2029-04-20 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  2-year progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
researchers who has been approved can share.